CLINICAL TRIAL: NCT00868816
Title: A Prospective, Randomized, Control Trial of Oxaliplatine Based Adjuvant Chemotherapy for Stage II/III Colorectal Cancer: 8 Cycles vs 12 Cycles
Brief Title: Oxaliplatine Based Adjuvant Chemotherapy for Stage II/III Colorectal Cancer: 8 Cycles Versus 12 Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: xu jianmin, zhongshan hospital, fudan university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Cancer
Keywords: oxaliplatine; colorectal cancer; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 12 cycles of oxaliplatine based adjuvant chemotherapy
  Interventions: Drug: 12 cycles of oxaliplatine based adjuvant chemotherapy
- 2 (Active Comparator): 8 cycles of oxaliplatine based adjuvant chemotherapy
  Interventions: Drug: 8 cycles of oxaliplatine based adjuvant chemotherapy

INTERVENTIONS:
Drug: 12 cycles of oxaliplatine based adjuvant chemotherapy — oxaliplatine 85 mg/㎡ d1, lv 200 mg/㎡ d1, 5-fu 1300 mg/㎡ ivgtt maintain for 48hr, every 3 weeks/cycle, 12 cycles
  Arms: 1
Drug: 8 cycles of oxaliplatine based adjuvant chemotherapy — oxaliplatine 85 mg/㎡ d1, lv 200mg/㎡ d1, 5-fu 1300 mg/㎡ ivgtt maintain for 48hr, every 3 weeks/cycle, 8 cycles
  Arms: 2

SUMMARY:
The purpose of this study is to investigate which oxaliplatie based adjuvant method (8 cycles or 12 cycles) is better for patients receiving curative colorectal cancer resection.

DETAILED DESCRIPTION:
We administered 5-FU, lv and Oxaliplatin as adjuvant chemotherapy (3 weeks per cycle) to patients with Stage II or Stage III colorectal cancer. The study endpoints were disease-free survival, overall survival, and liver metastasis-free survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age < 75 years with histologically proven adenocarcinoma of the colon or rectum
* no severe major organ dysfunction
* WHO performance status of 0 or 1
* Stage II (T3-4, N0, M0) or Stage III (T0-4, N1-2, M0) disease (according to the 1997 revision of the International Union Against Cancer TNM staging system)

Exclusion Criteria:

* age >= 75
* severe major organ dysfunction
* WHO performance status of >1
* Stage I or Stage IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 years after operation

SECONDARY OUTCOMES:
overall survival liver metastasis-free survival | 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, PHD, Study Director — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China